CLINICAL TRIAL: NCT06592534
Title: Babies With Enterocolitis - A Study of Faecal Calprotectin in Hirschsprung Disease (The BEACH Study)
Acronym: BEACH
Status: Not yet recruiting | Type: Observational
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Collaborators: Bowel Research UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 336089
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hirschprung's Disease; Hirschsprung Disease; Hirschsprung's Disease Associated Enterocolitis
Keywords: Faecal Calprotectin; Enterocolitis
MeSH Terms: conditions — Hirschsprung Disease; Enterocolitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants and children with Hirschsprung's Disease: Children under the age of 7 years with Hirschsprung's Disease.

SUMMARY:
Babies with Hirschsprung's Disease are born without normal nerves to the end of their bowel which means they cannot poo properly, and are at high risk of infection of the bowel, called enterocolitis. 1 in 4 children with Hirschsprung's Disease develop enterocolitis and, if not treated quickly, it can lead to death. The symptoms include a swollen tummy, temperatures and diarrhoea but it can be hard to spot, especially in the early stages, and there is no test for it.

In some diseases, a substance called calprotectin is found in the poo when the bowel is inflamed. The investigators plan to collect poo samples from children with Hirschsprung's Disease and measure the calprotectin, to see if it can help the investigators predict which children are at highest risk of enterocolitis. When the investigators collect the poo we will ask parents some questions about their child's diet and poos over the week before, and how easy it was to collect the sample.

This is a pilot study, which means the investigators don't expect to get a definite answer to whether measuring calprotectin levels will change treatment for children with Hirschsprung's disease. However, it will help the investigators find out if calprotectin levels are a useful test for bowel inflammation in these children and will tell us what parents' views are on collecting poo samples regularly. If it does look like measuring calprotectin is a useful test in Hirschsprung's disease, the investigators will do more studies to find out if some children may benefit from more intensive treatment.

DETAILED DESCRIPTION:
Background:

Hirschsprung's Disease is a rare congenital condition affecting 1 in 5000 children and characterised by an absence of ganglia in the distal bowel(1). Affected infants cannot stool normally and require an intensive treatment programme of regular rectal washouts or a stoma to ensure that their bowel is emptied, and avoid bowel perforation. Once they are a few months old definitive surgery is performed to remove the affected segment of bowel.

Infants with Hirschsprung's Disease have a high (1 in 4) risk of developing Hirschsprung's associated enterocolitis (HAEC), an inflammatory and infective condition of the bowel which can cause severe acute illness and death in 1-10% of affected children(2). Although the incidence of HAEC is reduced by surgery, the risk persists throughout childhood(3). Signs and symptoms are non-specific, including fevers, irritability, poor feeding, abdominal distension and explosive stool, and deterioration can be rapid. The mainstay of treatment is intravenous antibiotic therapy with colonic lavage per rectum. In severe cases, emergency surgery to remove the affected bowel is required, with long term implications for continence. A biomarker to identify children at higher risk of HAEC or its life-threatening complications would enable clinicians to consider employing additional or earlier treatments for these patients.

Faecal calprotectin is a biomarker currently used in both the diagnostic work-up of inflammatory bowel disease (IBD) and to monitor disease progression and remission, adding to the clinical decision making around escalation and de-escalation of IBD treatments(4, 5). Previous studies have demonstrated that faecal calprotectin levels reduce with age and have wide variability in early infancy(6).

Faecal calprotectin has not previously been described as a marker of enterocolitis in infants with Hirschsprung's Disease. We have received written communication of an unpublished retrospective study of single faecal calprotectin measurement in children with Hirschsprung's Disease and suspected HAEC from a UK centre. Using clinical, radiological, haematological and biochemical features this study divided 27 children into "low risk" and "high risk" groups. Faecal calprotectin level was significantly higher in the high risk group (285μg/g) compared to the low risk group (70μg/g) (p <0.01). Whilst these data suggest a potential role for faecal calprotectin assay in the diagnosis of acute HAEC, the difference might simply represent association due to demographics: baseline faecal calprotectin is known to be higher in younger children, likewise HAEC is more common in younger children with Hirschsprung's Disease. Further, it is unknown whether the 'high risk' group had a more profound acute calprotectin rise reflective of acute disease severity or a higher baseline. Serial faecal calprotectin monitoring could benefit children both for earlier diagnosis and earlier initiation of more intensive therapies.

Aim:

This study aims to describe the longitudinal changes observed in faecal calprotectin levels in infants and children with Hirschsprung's Disease. This pilot study will also be used to determine the acceptability of regular faecal calprotectin monitoring for parents using published and accepted methods(7) and will be used to power future studies.

Design:

This is a pragmatic research pilot study. Children under 5 years of age with biopsy proven Hirschsprung's Disease will be identified by the clinical team and invited to participate. Stool samples will be requested to be provided at every routine clinic appointment and elective admission and during any emergency admissions over the two year study period. The faecal calprotectin level will be analysed using standard laboratory protocols for each sample. At the time of each stool sample parents will be given a short questionnaire regarding the acceptability of collecting a stool sample and regarding their child's diet, bowel habits and recent illnesses.

The study will run for 2 years in 4 UK centres with an expectation that each patient provides a minimum of 4 samples to the study during this time. A control population has not been included as previous studies have shown that there is a very wide variability in faecal calprotectin in normal infants.

Descriptive analyses of the findings will be undertaken including analysis of the change in faecal calprotectin level over time including describing any changes associated with changes in diet; association with the number of episodes of HAEC; and the faecal calprotectin level at the time of admission with HAEC compared to the baseline level.

Key goals:

To describe the change in faecal calprotectin in early childhood of children with Hirschsprung's Disease An understanding of how an individual's faecal calprotectin levels change during infancy has not previously been described, particularly in children with Hirschsprung's Disease. This study will enable the investigators to track the faecal calprotectin levels over two years and to collect preliminary data to assess whether changes in diet and stooling patterns are associated with changes in faecal calprotectin.

To gain preliminary data to assess whether there may be an associated between faecal calprotectin and frequency or severity of HAEC episodes in young children with enterocolitis This pilot study will enable the investigators to undertake an initial assessment of whether there is any association between faecal calprotectin levels and HAEC and whether there is any association between faecal calprotectin level and severity of HAEC during an emergency admission.

To assess the acceptability to parents of taking stool samples regularly It is important to understand whether this is an acceptable sample to be collected by parents. Therefore, evaluating the acceptability of collecting a stool sample within the study will help the investigators to determine whether monitoring of faecal calprotectin levels would be possible within clinical practice. Children with Hirschsprung's Disease frequently stool with additional help, either through using rectal therapy or into a stoma bag, and therefore extrapolating the acceptability from people who do not have stooling difficulties is not appropriate.

Outcomes:

The results of this study will be presented in an international conference and will be published in a peer reviewed journal. The findings of this study are intended to determine whether faecal calprotectin has the potential to be used as a predictive biomarker for enterocolitis. If it is, we plan to undertake a definitive study to demonstrate this, using this study to power the sample size required. If faecal calprotectin proves a useful biomarker for determining the risk or severity of HAEC this will have important implications for patients, enabling them to be treated more intensively and effectively. Faecal calprotectin levels could also be used within the design of studies considering the efficacy of novel treatments of HAEC, as a recruitment criteria or as a method of stratifying HAEC severity.

ELIGIBILITY:
Inclusion criteria:

- Any infant or child under the age of 5 years at the time of recruitment with biopsy proven Hirschsprung's Disease

Exclusion criteria:

* Infants or children who do not have biopsy proven Hirschsprung's Disease
* Individuals with total colonic Hirschsprung's Disease
* Individuals with Hirschsprung's Disease which affects the small bowel
* Children aged 5 years and over at the time of recruitment
* Children with inflammatory bowel disease

Ages: 0 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and children will be identified during any admission to hospital, pre-operatively and during outpatient attendances.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Description of the change in baseline faecal calprotectin in infants with HSCR over time | 2 years
  This is a pilot study which aims to describe the baseline measurements and longitudinal changes observed in faecal calprotectin levels in children under the age of 7 years with Hirschsprung's Disease.

SECONDARY OUTCOMES:
Acceptability of repeated stool sampling | 2 years
  Validated questionnaire to determine the acceptability of repeated stool sampling. A score of 1 to 5 is given where 1 indicates poor acceptability and 5 indicates very good acceptance in each domain.

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised IPD will be shared upon reasonable request